CLINICAL TRIAL: NCT05809128
Title: Multidisciplinary Approach to Breast Cancer Through the Study of Altered Transcriptomic and Immune Accompanied by the Identification of Extractable Markers From the Radiodiagnostic Bioimaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS SYNLAB SDN (Other)
Responsible Party: Sponsor
Other Study IDs: 3/19
Record Dates: First submitted 2023-03-03; First posted 2023-04-12 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer Patients
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: surgery for breast cancer and imaging test evaluations — At the time of surgery, having completed the evaluation extemporaneous of the surgical piece, tissue samples will be collected to be stored from the material exceeding the completion of the patients' diagnosis. In addition, paramenters that can be extracted from radiodiagnostic images will be evaluated

SUMMARY:
Prospective observational study for onco-immunologic characterization and by bioimaging of breast neoplastic tissue of patients operated for breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of breast cancer.
* patients 25 to 80 years of age

Exclusion Criteria:

* Patients who refuse to participate in the study;
* Patients who do not fall within the age range mentioned above

Ages: 25 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Multiparametric flow cytometry analyses of Custer of Differentiation (CD) proteins expression on tumor infiltrating lymphocytes | 1-24 months
  The following phase of the study aims to go to evaluate the immunology of breast cancer patients compared with the control. In particular we will perfome an accurate characterization in flow cytometry of the cells present in the peripheral blood and of the immune component infiltrating the tumor (tumor infiltrating lymphocytes). The different components of tumor infiltrating lymphocytes will be assessed using the following antibodies: CD45 , CD8, CD4,CD3, HLA-DR, CD19 , CD 326 (EpCAM) ,CD56 , CD14 and CD16.
Analysis of gene expression profiles of cancer cells | 1-24 months
  The following area of study is focused on the study by molecular biology of samples of cancerous and healthy tissue that will be possible to obtain from the subjects participating in the study. For that phase, the type of instrumentation will be determined according to the amount of nucleic acids extracted from the tissues. In fact, samples that will allow recovery of high amounts of RNA and with a good degree of purity will be able to be used for studies carried out with next generation sequencing such as, for example, Ion Torrent S5. In the case of samples in which the RNA is difficult to extract or of low quality, methods such as real time polymerase chain reaction (PCR) in multiplex mode
Extraction of features from radiological images to be used as biomarkers. | 1-36 months
  Radiological images from High-field MRI, multilayer CT, hybrid systems such as PET-CT and PET-MRI will be use to extract quantitative parameters of the lesion and the other structures of interest. An automatic segmentation , or alternatively, a manual segmentation by an experienced radiologist or experienced nuclear physician will be performe.
Bioinformatics analysis | 37-48 months
  The correlations between the cytofluorimetric characterization of TILs and the quantitative parameters extracted from radiological images will be performed using different software such as Graphpad or ER softwares.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Synlab SDN, Naples, Italy